CLINICAL TRIAL: NCT00111592
Title: Effectiveness of a Treatment Protocol for Lower Urinary Tract Symptoms in General Practice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Yamanouchi (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MEC 00-007
Record Dates: First submitted 2005-05-23; First posted 2005-05-24 (Estimated); Last update posted 2016-11-09 (Estimated); Status verified 2007-11

CONDITIONS: Benign Prostatic Hyperplasia; Lower Urinary Tract Symptoms
Keywords: BPH; benign prostatic hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms | interventions — Clinical Protocols; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): current usual care
  Interventions: Procedure: current usual care
- 2 (Experimental): treatment protocol with clear indications for therapy
  Interventions: Procedure: treatment protocol with clear indications for therapy

INTERVENTIONS:
Procedure: current usual care — current usual care
  Arms: 1
Procedure: treatment protocol with clear indications for therapy — treatment protocol with clear indications for therapy
  Arms: 2

SUMMARY:
Ageing and the availability of medication has led to an increase of elderly male patients being treated for lower urinary tract symptoms (LUTS), or voiding problems ("prostate problems"). However, guidelines are vague as to which patients should and which should not be treated, and how.

Although several treatment modalities have proven efficacy in selected populations, it is unclear how effective these treatments are in daily practice.

This study investigates the hypothesis that a treatment protocol in which clear indications are formulated for all treatment modalities is more effective, as compared to current usual primary care, in reducing both symptoms as related to the quality of voiding in elderly males.

DETAILED DESCRIPTION:
Guidelines fail to provide specific diagnostic criteria and clear indications for therapy in elderly male patients with lower urinary tract symptoms. Consequently, the group of patients diagnosed with LUTS in primary care is very heterogeneous, and daily care varies widely.

Consequently, efficacy trials of alpha-blockers, 5-alpha-reductase inhibitors and surgery performed in selected, well defined homogeneous populations cannot easily be generalised to the heterogeneous primary care situation.

A practical randomised trial enrolling patients on the basis of symptoms have the advantage of being of immediate practical value.

We compare a treatment protocol with clear indications for therapy with current usual care in a population selected on symptoms rather than well defined diseases or definite test results.

Two hundred eight subjects were randomised into intervention (N=104) and control (N=104) conditions.

After two years of follow-up, IPSS scores, bother scores, maximum urinary flow rates and the incidence of acute urinary retention and urinary tract infections have been compared.

ELIGIBILITY:
Inclusion Criteria:

* International Prostate Symptom Score > 7
* Age > 55 years

Exclusion Criteria:

* Heart failure
* Diabetes type I
* Psychiatric disorder/cognitive dysfunction
* History of prostate surgery
* Active treatment for lower urinary tract symptoms

Min Age: 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2000-08; Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Degree of lower urinary tract symptoms (International Prostate Symptom Score [IPSS])
Maximum urinary flow rate (Qmax)

SECONDARY OUTCOMES:
Bother due to lower urinary tract symptoms (Danish-Prostatic Symptom Score [Dan-PSS])
incidence of acute urinary retention
incidence of urinary tract infections

CONTACTS AND LOCATIONS:
Overall Officials: Roelf Norg, Principal Investigator — Department of General Practice, Universiteit Maastricht
Locations (1):
- University of Maastricht, Department of General Practice, Maastricht, Limburg, Netherlands